CLINICAL TRIAL: NCT03474913
Title: Feasibility and Efficacy of Upright MP - MRI for Prostate Cancer Screening
Brief Title: Upright MRI for Prostate Cancer Screening
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: The Fonar Corporation (Unknown)
Responsible Party: Principal Investigator, Ashutosh Kumar Tewari, Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 17-2776
Record Dates: First submitted 2018-03-16; First posted 2018-03-23 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Elevated PSA; Elevated Prostate Specific Antigen
Keywords: Prostate Cancer Diagnosis; Imaging; Magnetic Resonance Imaging; Cancer; Diagnostic; Malignant Neoplasm of Prostate
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Prostate Biopsy Cores and/or Punch Cores from Radical Prostatectomy Specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Standard MRI first: Patients will have a standard of care MRI, then consent to study participation and have an upright MRI.
  Interventions: Device: Upright MRI
- MRIs in random order: Patients will consent to participate in the study, then do two MRIs in random order.
  Interventions: Device: Upright MRI; Device: Standard MRI

INTERVENTIONS:
Device: Upright MRI — Indomitable Magnetic Resonance Imaging Scanner, magnetic resonance imaging using 0.6 T strength
Device: Standard MRI — standard of care closed 3T MRI
  Groups: MRIs in random order

SUMMARY:
This is an investigator initiated study to test the efficacy of an upright MRI (Magnetic Resonance Imaging) for the screening of prostate cancer. The purpose of this study is to compare Upright MRI as a technique to PSA (Prostate Specific Antigen) and current MRI imaging. It will take place at Mount Sinai Hospital, and last for a total of about 5 years. Eligible patients will be determined by the urologist. The target population is men who are at risk for prostate cancer, as determined by the urologist. Diagnostic criteria will include elevated PSA and an abnormal digital rectal exam (DRE). After patients are screened and determined eligible, they will be asked to have a seated MRI using the Indomitable Magnetic Resonance Imaging Scanner, Ex vivo magnetic resonance imaging using 0.6 T strength, as well as a standard of care closed 3T MRI. After each scan, the patient will be given a series of questionnaires to assess their comfort level during the scan. Patients will be followed every 6 months after completion of (or early withdrawal from) study enrollment until 5 years.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the second most common cancer among men in the United States, with over 180,000 new cases diagnosed in 2016. This commonality implies that set standards need to be set and devise effective tools to screen and diagnose prostate cancer. Today, prostate specific antigen (PSA) test is the most widely adopted screening method for PCa. Since its introduction in 1979, it has helped in earlier diagnosis of PCa and has had a marked shift on the stage at which PCa is identified. PSA, although popular as a screening tool, has several shortcomings. It is organ-specific rather than cancer-specific, which means that its values can be elevated even for non-malignant conditions . Indeed, PSA based screening has reported positive predictive value as low as 30% (PSA cutoff >4.0 ng/dL) for detecting prostate cancer and an over diagnosis rate of 50%, which leads to unnecessary biopsies and aggressive treatments of men with clinically indolent (insignificant) disease.

Current diagnostic pathway of prostate cancer requires men with elevated PSA and abnormal Digital Rectal exam to undergo a Trans Rectal Ultra Sound (TRUS) guided biopsy. TRUS is a blind-systematic biopsy, which randomly samples prostate tissue. This can lead to missing or under-diagnosing clinically significant cancer and over-diagnosing clinically insignificant disease. TRUS biopsy is itself associated with morbidity, mainly in the form of hematuria, hematospermia, pain, urinary retention and sometimes can cause life-threatening sepsis.

Many of the PSA screened detected prostate cancers detected on TRUS are clinically insignificant and even if left untreated have little to no clinical impact on an individual's remaining life. Overtreatment resulting from over diagnosis often leads to side effects like erectile dysfunction (approx. 60%) from radical therapy and urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Men at risk of prostate cancer and have been advised to have a prostate MRI.
* Age ≥ 18 years.
* Fit for undergoing all study protocol procedures which includes an ultrasound guided biopsy.
* Able to tolerate general or spinal anesthesia.
* Ability to understand and the willingness to sign a written informed consent and to comply with the protocol.

Exclusion Criteria:

* Patients who have been treated using 5- alpha-reductase inhibitors at the time of study enrollment or 6 months prior to enrollment.
* Patients with previous history of prostate biopsy, prostate surgery or treatment for prostate cancer (interventions for benign prostatic hyperplasia/bladder outflow obstruction is acceptable)
* Patients who have evidence of a urinary tract infection or history of acute prostatitis within the last 3 months.
* Patients contraindicated to undergoing the MRI procedure e.g. pacemaker, estimated GFR<=50, automatic implantable cardiac defibrillators.
* History of any other medical condition precluding procedures described in the protocol

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women do not have prostates and this is a study of prostate health
Study Population: Men at risk for prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
PSA levels | 5 years
  Prostate-specific Antigen (PSA) levels

SECONDARY OUTCOMES:
Upright MRI compared to Standard MRI | 5 years
  To compare performance characteristics of Upright MP-MRI versus 3T MP-MRI in detecting clinically significant PCa and PCa in general.
Claustrophobic Questionnaire (CLQ) | 5 years
  Claustrophobic Questionnaire (CLQ) is a 46 item instrument, each item score on a likert scale from 1-5, full scale from 36 to 180, with higher score indicating more anxiety.
NCCN Distress Thermometer | 5 years
  NCCN Distress Thermometer is a visual scale - full scale from 0-10, higher score indicating higher level of distress
Magnetic Resonance Imaging-Anxiety Questionnaire (MRI-AQ) | 5 years
  Magnetic Resonance Imaging-Anxiety Questionnaire (MRI-AQ) is a 15 item instrument, each item score on a likert scale from 1 to 4, full scale range from 15 to 66, with higher score indicating higher degree of anxiety.
Diagnostic Yield of MRI and PSA Density | 5 years
  To compare the diagnostic yield of using MP-MRI with thresholds PSA density used for detecting prostate cancer.
Number of Correctly Identified side | 5 years
  Number of correctly identified side of prostate unaffected in men with pathological disease

CONTACTS AND LOCATIONS:
Overall Officials: Ash Tewari, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided